CLINICAL TRIAL: NCT00005044
Title: A Phase III Trial to Evaluate the Duration of Neoadjuvant Total Androgen Suppression (TAS) and Radiation Therapy (RT) in Intermediate-Risk Prostate Cancer
Brief Title: Hormone Therapy and Radiation Therapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-9910; CDR0000067635
Record Dates: First submitted 2000-04-06; First posted 2003-01-27 (Estimated); Results first posted 2017-10-31 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-05

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Flutamide; Gonadotropin-Releasing Hormone; Goserelin; Leuprolide; luprolide acetate gel depot; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAS x 8 weeks (Experimental): Total Androgen Suppression (TAS) (LHRH agonist and Casodex or Eulexin) x 8 weeks followed by radiation therapy (RT) with concurrent TAS (LHRH agonist and Casodex or Eulexin).
  Interventions: Drug: Casodex; Drug: Eulexin; Drug: LHRH agonist; Radiation: radiation therapy
- TAS x 28 weeks (Experimental): TAS (LHRH agonist and Casodex or Eulexin) x 28 weeks followed by RT with concurrent TAS (LHRH agonist and Casodex or Eulexin).
  Interventions: Drug: Casodex; Drug: Eulexin; Drug: LHRH agonist; Radiation: radiation therapy

INTERVENTIONS:
Drug: Casodex — Orally at a dose of one 50 mg tablet per day started within (before or after) 14 days of the first LHRH agonist injection.
  Other Names: bicalutamide
Drug: Eulexin — Orally at a dose of two 125 mg capsules three times a day for a total daily dose of 750 mg (six capsules) started within (before or after) 14 days of the first LHRH agonist injection.
  Other Names: flutamide
Drug: LHRH agonist — LHRH agonist of choice. The manufacturer's instructions should be followed.
  Other Names: Zoladex; Lupron; Eligard; Viadur; luteinizing hormone-releasing hormone (LHRH)-agonist
Radiation: radiation therapy — [Prostate and any extraprostatic tumor extension + 1.0-1.5 cm margin receives 70.2 Gy (1.8 Gy/day x 39 fractions, five days/week)] OR [regional nodes, prostate and seminal vesicles + 1.0-1.5 cm margin will receive 46.8 Gy (1.8 Gy/day x 26 fractions, five days/week), followed by a 23.4 Gy (1.8 Gy/day x 13 fractions, five days/week) boost to the prostate and any extraprostatic tumor extension + 1.0-1.5 cm margin]

SUMMARY:
RATIONALE: Hormones can stimulate the growth of prostate cancer cells. Hormone therapy may fight prostate cancer by reducing the production of androgens. Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known which regimen of hormone therapy and radiation therapy is more effective for prostate cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of two different regimens of hormone therapy and radiation therapy in treating patients who have prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of moderate-duration (28 weeks) neoadjuvant total androgen suppression (TAS) and radiotherapy (RT) with short-duration (8 weeks) neoadjuvant TAS and RT, as related to disease-specific survival, in patients with intermediate-risk adenocarcinoma of the prostate.
* Compare these regimens, in terms of overall survival, disease-free survival, time to local tumor progression or distant failure, time to first biochemical failure, hormone-refractory state, and treatment-induced morbidity, in this patient population.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to prostate-specific antigen level (no greater than 10 ng/mL vs greater than 10 but no greater than 20 ng/mL vs greater than 20 ng/mL), tumor stage (T1b-2 vs T3-4), Gleason score (2-4 vs 5-6 vs 7-10), and prior hormonal therapy (yes vs no). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive total androgen suppression for 8 weeks prior to the initiation of radiotherapy and throughout radiotherapy. A luteinizing hormone-releasing hormone (LHRH) agonist is administered every 1-3 months AND bicalutamide OR flutamide is given orally daily for a total duration of 16 weeks. Beginning with week 9, patients undergo radiotherapy 5 days a week for 8 weeks.
* Arm II: Patients receive total androgen suppression for 28 weeks prior to the initiation of radiotherapy and throughout radiotherapy. An LHRH agonist AND bicalutamide OR flutamide are administered as in arm I for a total duration of 36 weeks. Beginning with week 29, patients undergo radiotherapy as in arm I.

Patients are followed every 3 months for 1 year, every 6 months for 4 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 1,540 patients (770 per treatment arm) will be accrued for this study within 4 years.

ELIGIBILITY:
Inclusion Criteria

1. Adenocarcinoma of prostatic origin histologically-confirmed within 180 days of the randomization date.
2. Zubrod Performance Status 0-1 (Appendix II).
3. Prostatic biopsy tumor grading by the Gleason Score classification (Appendix VI) is mandatory prior to randomization.
4. Patients at intermediate risk for disease relapse as determined by any of the following combinations of factors (NOTE: tumor found in one or both lobes on biopsy, but not palpable, will not alter T stage):

   * Clinical stage T1b-4, Gleason score 2-6, and prostate-specific antigen >10 but ≤ 100.
   * Clinical stage T1b-4, Gleason score 7, and prostate-specific antigen < 20.
   * Clinical stage T1b-1c, Gleason score 8-10, and prostate-specific antigen <20.
5. Clinically negative (N0) lymph nodes (LN) as established by imaging (pelvic ± abdominal CT, MRI or LAG), or negative LN by nodal sampling or dissection (laparoscopy or laparotomy). Patients with radiologic (e.g., CT, MRI or LAG) or radioimmunoscintigraphy (i.e., ProstaScint™) findings suggestive of regional nodal involvement are eligible if cytologic (e.g., needle aspiration) or histologic (e.g., surgical sampling) evaluation shows no evidence of a neoplastic process (i.e., prostatic or non-prostatic malignancy). Patients with equivocal radiologic findings (maximum nodal size ≤ 1.5 cm) are eligible.
6. No distant (M0) metastases. Patients with radionuclide imaging (e.g., bone scintigraphy, ProstaScint™) findings suggestive, but not diagnostic of metastatic disease are eligible if radiologic (e.g., standard or tomographic radiography, or CT/MRI) imaging does not confirm metastatic disease.
7. Pretherapy serum (total) prostate-specific antigen value performed with a Federal Drug Administration approved assay method, e.g. Abbott, Hybritech, etc.
8. Treatment must begin within 6 weeks after randomization.
9. Alanine aminotransferase (ALT) must be within 2 x upper normal limit.
10. Patients must sign a study-specific informed consent form (Appendix I) prior to randomization.

Exclusion Criteria

1. Patients at high risk for disease relapse as determined by either:

   * Prostate-specific antigen ≥ 20 and Gleason score ≥ 7 (any T stage).
   * Clinical stage ≥T2 and Gleason score ≥ 8 (any prostate-specific antigen).
2. Patients at low risk for disease relapse as determined by:

   • Clinical stage ≤T2, Gleason score ≤ 6, and prostate-specific antigen ≤ 10.
3. Clinical stage Tx, T0, or T1a.
4. Histologic or radiologic evidence of tumor involvement of regional lymph nodes (N1) or the presence of metastatic disease (M1).
5. Pretherapy serum prostate-specific antigen level > 100.
6. Co-morbid medical illness which in the opinion of the investigator is expected to result in a life expectancy of <10 years.
7. Any of the following prior therapies:

   * Pelvic external beam radiation therapy.
   * Radionuclide prostate brachytherapy.
   * Prostatectomy or prostatic cryosurgery.
   * Prior bilateral orchiectomy.
   * Prior androgen suppression therapy; however, patients begun on LHRH agonist therapy remain eligible if (1) LHRH agonists were started no more than 30 days before randomization, and (2) Casodex or Eulexin was (or will be) started no more than 14 days before or after the date that the LHRH agonist injection was given. Any finasteride therapy administered for prostatic hypertrophy must be discontinued.
   * Chemotherapy for prostatic carcinoma.
8. Previous or concomitant invasive cancer, other than localized basal cell or squamous cell skin carcinoma (AJCC Stage 0-II), unless continually disease free for at least 5 years.
9. Major medical or psychiatric illness which, in the opinion of the investigator, would prevent completion of treatment or would interfere with follow-up.
10. The patient's participation in another medical research study that involves prostate cancer treatment.

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1579 (Actual)
Dates: Start 2000-02 (Actual); Primary Completion 2012-09 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael G. Haddock, MD, Study Chair — Mayo Clinic
Locations (261):
- United States (241):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Comprehensive Cancer Institute, Huntsville, Alabama
  - Huntsville Hospital, Huntsville, Alabama
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - Montgomery Cancer Center, Montgomery, Alabama
  - DCH Cancer Treatment Center, Tuscaloosa, Alabama
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Mount Diablo Medical Center, Concord, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - California Cancer Center, Fresno, California
  - Saint Agnes Cancer Center, Fresno, California
  - Sutter Health Western Division Cancer Research Group, Greenbrae, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Huntington Cancer Center at Huntington Hospital, Pasadena, California
  - Robert and Beverly Lewis Family Cancer Care Center, Pomona, California
  - Radiation Oncology Center - Sacramento, Sacramento, California
  - Radiation Medical Group, Incorporated, San Diego, California
  - Naval Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - O'Connor Hospital, San Jose, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Torrance Memorial Medical Center, Torrance, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - Hospital of St. Raphael, New Haven, Connecticut
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - 21st Century Oncology - Fort Myers, Fort Myers, Florida
  - Shands Cancer Center at the University of Florida Health Science Center, Gainesville, Florida
  - Florida Radiation Oncology Group, Jacksonville, Florida
  - Holmes Regional Medical Center, Melbourne, Florida
  - University of Miami Sylvester Cancer Center, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Bay Medical Center, Panama City, Florida
  - Gulf Coast Cancer Treatment Center, Panama City, Florida
  - Sarasota Radiation and Medical Oncology Center, Sarasota, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Medical Center/John B. Amos Community Cancer Center, Columbus, Georgia
  - Regional Radiation Oncology Center at Rome, Rome, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - CCOP - Scott and White Hospital, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - St. John's Medical Center, Anderson, Indiana
  - Bloomington Hospital, Bloomington, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - Methodist Cancer Center at Methodist Hospital, Indianapolis, Indiana
  - Community Regional Cancer Care, Indianapolis, Indiana
  - Ball Memorial Hospital Cancer Center, Muncie, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Wendt Regional Cancer Center of Finley Hospital, Dubuque, Iowa
  - St. Elizabeth Medical Center, Edgewood, Kentucky
  - Central Baptist Hospital, Lexington, Kentucky
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Louisville Radiation Oncology Center at Caritas Regional Cancer Center, Louisville, Kentucky
  - Merle M. Mahr Cancer Center, Madisonville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Anne Arundel Oncology Center, Annapolis, Maryland
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Greater Baltimore Medical Center and Cancer Center, Baltimore, Maryland
  - Harbor Hospital Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - St. Agnes Cancer Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - NSMC Cancer Center, Peabody, Massachusetts
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - McLaren Regional Cancer Center, Flint, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Marquette General Hospital, Marquette, Michigan
  - MidMichigan Medical Center - Midland, Midland, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - William Beaumont Hospital - Royal Oak, Royal Oak, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Fairview University Medical Center - University Campus, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Hospital Cancer Center, St Louis, Missouri
  - Mallinckrodt Institute of Radiology, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Hospital Cancer Center at Nebraska Methodist Hospital - Omaha, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth Medical School, Lebanon, New Hampshire
  - Elliot Regional Cancer Center, Manchester, New Hampshire
  - Cooper Cancer Institute, Camden, New Jersey
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - John F. Kennedy Medical Center, Edison, New Jersey
  - Trinitas Hospital - Jersey Street Campus, Elizabeth, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - South Jersey Regional Cancer Center, Millville, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital, Mount Holly, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Atlantic City Medical Center, Pomona, New Jersey
  - Medical Center of Princeton, Princeton, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Somerset Medical Center, Somerville, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Fox Chase Cancer Center at St. Francis Medical Center, Trenton, New Jersey
  - Associated Radiologists, P.A., Warren Township, New Jersey
  - Radiation Oncology Associates of Albuquerque, Albuquerque, New Mexico
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Finger Lakes Radiation Oncology Center, Clifton Springs, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Beth Israel Medical Center - Philipps Ambulatory Care Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Riverhill Radiation Oncology, Yonkers, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Batte Cancer Center at Northeast Medical Center, Concord, North Carolina
  - Leo W. Jenkins Cancer Center of University Health Systems of Eastern Carolina, Greenville, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Trinity Cancer Care Center, Minot, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Akron City Hospital, Akron, Ohio
  - Cancer Center at Christ Hospital, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Parma Community General Hospital, Parma, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Frank C. Love Cancer Institute at St. Anthony Hospital, Oklahoma City, Oklahoma
  - Oklahoma University Medical Center at University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - St. John Health System, Tulsa, Oklahoma
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - John and Dorothy Morgan Cancer Center at Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke's Hospital Cancer Center, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Pocono Cancer Center, East Stroudsburg, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Abramson Cancer Center at University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Veterans Affairs Medical Center - Philadelphia, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Mercy Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Wilkes-Barre General Hospital, Wilkes-Barre, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Wellspan Health - York Cancer Center, York, Pennsylvania
  - Roger Williams Medical Center, Providence, Rhode Island
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - West Tennessee Cancer Center at Jackson-Madison County General Hospital, Jackson, Tennessee
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Arlington Cancer Center, Arlington, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Bayshore Medical Center, Pasadena, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - Green Mountain Oncology Group, Bennington, Vermont
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - RMH Regional Cancer Center, Harrisonburg, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Bon Secours - St. Mary's Hospital, Richmond, Virginia
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - Cancer Institute at Virginia Mason Medical Center, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Yakima Valley Memorial Hospital, Yakima, Washington
  - Schiffler Cancer Center, Wheeling, West Virginia
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Southern Wisconsin Radiotherapy Center, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - Columbia Hospital, Milwaukee, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
  - All Saints Cancer Center at All Saints Healthcare, Racine, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
- Canada (20):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Doctor Leon Richard Oncology Centre, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre - Sudbury, Greater Sudbury, Ontario
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Northwestern Ontario Regional Cancer Care, Thunder Bay, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Result] Pisansky TM, Hunt D, Gomella LG, Amin MB, Balogh AG, Chinn DM, Seider MJ, Duclos M, Rosenthal SA, Bauman GS, Gore EM, Rotman MZ, Lukka HR, Shipley WU, Dignam JJ, Sandler HM. Duration of androgen suppression before radiotherapy for localized prostate cancer: radiation therapy oncology group randomized clinical trial 9910. J Clin Oncol. 2015 Feb 1;33(4):332-9. doi: 10.1200/JCO.2014.58.0662. Epub 2014 Dec 22. PMID 25534388
- [Derived] Spratt DE, Tang S, Sun Y, Huang HC, Chen E, Mohamad O, Armstrong AJ, Tward JD, Nguyen PL, Lang JM, Zhang J, Mitani A, Simko JP, DeVries S, van der Wal D, Pinckaers H, Monson JM, Campbell HA, Wallace J, Ferguson MJ, Bahary JP, Schaeffer EM, Sandler HM, Tran PT, Rodgers JP, Esteva A, Yamashita R, Feng FY. Artificial Intelligence Predictive Model for Hormone Therapy Use in Prostate Cancer. NEJM Evid. 2023 Aug;2(8):EVIDoa2300023. doi: 10.1056/EVIDoa2300023. Epub 2023 Jun 29. PMID 38320143

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TAS x 8 Weeks | TAS x 28 Weeks
Started | 790 | 789
Completed | 752 (Subjects with data available for the primary analysis are considered to have completed the study.) | 737 (Subjects with data available for the primary analysis are considered to have completed the study.)
Not Completed | 38 | 52
Not completed — Protocol Violation | 37 | 46
Not completed — Withdrawal by Subject | 1 | 5
Not completed — No protocol treatment | 0 | 1

BASELINE CHARACTERISTICS:
Population: Eligible patients with follow-up data
Groups:
- Total: Total of all reporting groups
Arm/Group | TAS x 8 Weeks | TAS x 28 Weeks | Total
Number analyzed (Participants) | 752 | 737 | 1489
Age, Continuous [Median (Full Range); unit: years] | 71 [45 to 84] | 71 [46 to 88] | 71 [45 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 752 | 737 | 1489

OUTCOME MEASURES:

1. Primary Outcome: Disease-specific Survival (DSS) (10-year Rates Reported)
Description: Disease-specific survival time is measured from date of randomization to death due to prostate cancer based on study chair review, with prostate-cancer death defined as (1) primary cause of death certified as due to prostate cancer, (2) complication of therapy, irrespective of disease status, (3) disease progression in the absence of any anti-tumor therapy, or (4) a 1.0 ng/ml-exceeding-rise in serum prostate-specific antigen (PSA) level on at least two consecutive occasions that occurs during or after salvage androgen suppression therapy. Death due to other causes is considered a competing risk. All others are censored. DSS is estimated using the cumulative incidence method. Ten-year rate is reported.
Time Frame: From randomization to 10 years. (Patients are followed until death or study termination, whichever occurs first.)
Population: Eligible patients with follow-up data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAS x 8 Weeks | TAS x 28 Weeks
Number analyzed (Participants) | 752 | 737
percentage of participants | 95 [93 to 97] | 96 [95 to 98]
Statistical Analysis 1: Comparison: TAS x 8 Weeks vs TAS x 28 Weeks; Assuming 40% of deaths in the 8-wk arm from prostate cancer (PC) and that 8-yr DSS would be 79%, 270 PC deaths were required to detect a 33% hazard reduction in the 28-wk arm with 90% power using the log-rank test with a 2-sided significance level of 0.05. Under assumed failure rates, 1,540 patients accrued over 4 years and observed for an additional 6 years were expected to provide the requisite events. This sample accounted for a 10% ineligible/lack-of-data rate and 3 interim analyses; Test type: Superiority; p = 0.45, Log Rank; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.48 to 1.39] — Reference level = TAS x 8 weeks

2. Secondary Outcome: Overall Survival (OS) (10-year Rates Reported)
Description: Survival time is defined as time from randomization to the date of death from any cause and is estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact. Ten-year rate is reported.
Time Frame: From randomization to 10 years. (Patients are followed until death or study termination, whichever occurs first.)
Population: Eligible patients with follow-up data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAS x 8 Weeks | TAS x 28 Weeks
Number analyzed (Participants) | 752 | 737
percentage of participants | 66 [62 to 70] | 67 [63 to 71]
Statistical Analysis 1: Comparison: TAS x 8 Weeks vs TAS x 28 Weeks; With 1540 patients accrued over 4 years and observed for an additional 6 years, determined for the primary endpoint, there would be 90% power to detect a 22% reduction in the hazard of all cause deaths in the 28-week arm, with 2-sided significance level of 0.05. This sample accounted for a 10% ineligible/lack-of-data rate; Test type: Superiority; p = 0.62, Log Rank; 2-sided significance level of 0.05; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.79 to 1.15] — Reference level = TAS x 8 weeks

3. Secondary Outcome: Disease-free Survival (DFS) (10-year Rates Reported)
Description: Disease-free survival time is defined as time from randomization to the date of disease progression or death from any cause and is estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact. Ten-year rate is reported.
Time Frame: From randomization to 10 years. (Patients are followed until death or study termination, whichever occurs first.)
Population: Eligible patients without follow-up data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAS x 8 Weeks | TAS x 28 Weeks
Number analyzed (Participants) | 752 | 737
percentage of participants | 24 [20 to 27] | 23 [20 to 27]
Statistical Analysis 1: Comparison: TAS x 8 Weeks vs TAS x 28 Weeks; Test type: Superiority; p = 0.47, Log Rank; Significance level = 0.05; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.85 to 1.08] — Reference level = TAS x 8 weeks

4. Secondary Outcome: Clinical Patterns of Tumor Recurrence: Time to Locoregional Progression (LRP) and Time to Distant Metastasis (DM) (10 Year Rates Reported)
Description: Time to distant metastasis measured from date of randomization to date of documented distant metastasis; competing risks are BF, LRP, and death without DM; all others are censored. Time to locoregional progression measured from date of randomization to date of documented local or regional progression; competing risks are BF [protocol definition- first of (1) the midway date between the last non-rising PSA and the first rising PSA of three consecutive rises or (2) the date of the initiation of salvage hormone therapy], DM, and death without LRP; all others are censored. LRP and DM are estimated using the cumulative incidence method. Ten -year rates are reported.
Time Frame: From randomization to 10 years. (Patients are followed until death or study termination, whichever occurs first.)
Population: Eligible patients with follow-up data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAS x 8 Weeks | TAS x 28 Weeks
Number analyzed (Participants) | 752 | 737
percentage of participants
  Locoregional progression | 6 [4 to 8] | 4 [3 to 6]
  Distant metastasis | 6 [4 to 8] | 6 [4 to 8]
Statistical Analysis 1: Comparison: TAS x 8 Weeks vs TAS x 28 Weeks; Locoregional progression; Test type: Superiority; p = 0.07, Gray's test; 2-sided significance level = 0.05; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.40 to 1.05] — Reference level = TAS x 8 weeks
Statistical Analysis 2: Comparison: TAS x 8 Weeks vs TAS x 28 Weeks; Distant metastasis; Test type: Superiority; p = 0.80, Gray's test; 2-sided significance level = 0.05; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.68 to 1.66] — Reference level = TAS x 8 weeks

5. Secondary Outcome: Time to First Biochemical Failure (BF) (10-year Rates Reported)
Description: Protocol definition: Time to BF measured from date of randomization to first of (1) the midway date between the last non-rising PSA and the first rising PSA of three consecutive rises or (2) the date of the initiation of salvage hormone therapy; competing risks are LRP, DM, and death without BF; all others are censored.
  Phoenix definition: Time to BF measured from date of randomization to first of (1) the date of documented rise of 2 ng/ml above the post-treatment(RT end date) nadir or (2) the date of the initiation of salvage hormone therapy; competing risks are LRP, DM, and death without BF; all others are censored. For both definitions BF is estimated using the cumulative incidence method. Ten year rates reported.
Time Frame: From randomization to 10 years. (Patients are followed until death or study termination, whichever occurs first.)
Population: Eligible patients with follow-up data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAS x 8 Weeks | TAS x 28 Weeks
Number analyzed (Participants) | 752 | 737
percentage of participants
  Protocol definition | 56 [52 to 59] | 59 [56 to 63]
  Phoenix definition | 27 [23 to 30] | 27 [23 to 30]
Statistical Analysis 1: Comparison: TAS x 8 Weeks vs TAS x 28 Weeks; Protocol definition; Test type: Superiority; p = 0.74, Gray's test; 2-sided significance level = 0.05; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.89 to 1.17] — Reference level = TAS x 8 weeks
Statistical Analysis 2: Comparison: TAS x 8 Weeks vs TAS x 28 Weeks; Phoenix definition; Test type: Superiority; p = 0.77, Gray's test; 2-sided significance level = 0.05; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.79 to 1.19] — Reference level = TAS x 8 weeks

6. Secondary Outcome: Time to Second Biochemical Failure (SBF) (10-year Rates Reported)
Description: Time to SBF measured from date of randomization to the date of PSA increase of ≥1.0 ng/mL (from the nadir PSA after completion of protocol-specified therapy) after salvage androgen suppression was started; competing risks LRP, DM, and death without SBF; all others are censored. SBF is estimated using the cumulative incidence method. Ten-year rates are reported.
Time Frame: From randomization to 10 years. (Patients are followed until death or study termination, whichever occurs first.)
Population: Eligible patients with follow-up data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAS x 8 Weeks | TAS x 28 Weeks
Number analyzed (Participants) | 752 | 737
percentage of participants | 10 [7 to 12] | 9 [7 to 12]
Statistical Analysis 1: Comparison: TAS x 8 Weeks vs TAS x 28 Weeks; Test type: Superiority; p = 0.62, Log Rank; 2-sided significance level = 0.05; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.64 to 1.30] — Reference level = TAS x 8 weeks

7. Secondary Outcome: Treatment-induced Morbidity (Highest Grade Toxicity Reported Per Patient)
Description: Acute drug therapy and radiation (<= 90 days from start of RT) toxicity was graded using the Common Toxicity Criteria (CTC) v.2.0 criteria; late toxicity was graded using the Radiation Therapy Oncology Group (RTOG)/European Organisation for Research and Treatment of Cancer (EORTC) Late Radiation Morbidity Scoring schema. Grade refers to the severity of the toxicity. The CTC v2.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each toxicity based on this general guideline: Grade 1 Mild toxicity, Grade 2 Moderate toxicity, Grade 3 Severe toxicity, Grade 4 Life-threatening or disabling toxicity, Grade 5 Death related to toxicity. The highest grade acute and late toxicity was determined for each patient.
Time Frame: From randomization to 10 years. (Patients are followed until death or study termination, whichever occurs first.)
Population: Eligible patients with adverse event data in corresponding time frame (during hormone therapy and <=90 days from RT start; > 90 days from RT start)
Measure: Number; unit: percentage of participants
Arm/Group | TAS x 8 Weeks | TAS x 28 Weeks
Number analyzed (Participants) | 747 | 735
percentage of participants
  Acute RT and Hormone Toxicity: Grade 1 | 30.8 | 19.5
  Acute RT and Hormone Toxicity: Grade 2 | 41.6 | 49.8
  Acute RT and Hormone Toxicity: Grade 3 | 16.1 | 25.7
  Acute RT and Hormone Toxicity: Grade 4 | 0 | 0.1
  Acute RT and Hormone Toxicity: Grade 5 | 0 | 0
  Late RT Toxicity: Grade 1: number analyzed (Participants) | 742 | 724
  Late RT Toxicity: Grade 1 | 34.0 | 32.9
  Late RT Toxicity: Grade 2: number analyzed (Participants) | 742 | 724
  Late RT Toxicity: Grade 2 | 20.5 | 22.5
  Late RT Toxicity: Grade 3: number analyzed (Participants) | 742 | 724
  Late RT Toxicity: Grade 3 | 9.7 | 8.0
  Late RT Toxicity: Grade 4: number analyzed (Participants) | 742 | 724
  Late RT Toxicity: Grade 4 | 0.1 | 0.3
  Late RT Toxicity: Grade 5: number analyzed (Participants) | 742 | 724
  Late RT Toxicity: Grade 5 | 0 | 0

ADVERSE EVENTS:
Description: Eligible patients with adverse event data are included. Subjects experiencing more than one of a given adverse event are counted only once for that adverse event.
Arm/Group | TAS x 8 Weeks | TAS x 28 Weeks
Serious Adverse Events (participants affected / at risk) | 121/747 | 109/735
Other Adverse Events (participants affected / at risk) | 695/747 | 707/735
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAS x 8 Weeks (N=747) | TAS x 28 Weeks (N=735)
Arrhythmia NOS (Cardiac disorders) | 1 | 0
Supraventricular arrhythmia NOS (Cardiac disorders) | 0 | 1
Diarrhea NOS (Gastrointestinal disorders) | 12 | 18
Gastritis NOS (Gastrointestinal disorders) | 0 | 1
Late RT Toxicity: Other GI: NOS (Gastrointestinal disorders) | 10 | 3
Late RT Toxicity: Small/Large Intestine: NOS (Gastrointestinal disorders) | 9 | 8
Proctalgia (Gastrointestinal disorders) | 0 | 1
Proctitis NOS (Gastrointestinal disorders) | 1 | 1
Vomiting NOS (Gastrointestinal disorders) | 1 | 0
Late RT Toxicity: Other: NOS (General disorders) | 24 | 26
Pain-other (General disorders) | 1 | 0
Hepatic-Other (Hepatobiliary disorders) | 0 | 1
Infection with unknown ANC (Infections and infestations) | 0 | 1
Infection, Other (Infections and infestations) | 0 | 1
Dermatitis radiation NOS (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 15 | 4
Aspartate aminotransferase increased (Investigations) | 4 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia NOS (Metabolism and nutrition disorders) | 2 | 3
Hypoglycaemia NOS (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Headache NOS (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 6 | 1
Late RT Toxicity: Bladder: NOS (Renal and urinary disorders) | 33 | 24
Renal/GU-Other (Renal and urinary disorders) | 1 | 2
Urinary retention (Renal and urinary disorders) | 1 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1
Late RT Toxicity: Other GU: NOS (Reproductive system and breast disorders) | 21 | 25
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea NOS (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary-other (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 0 | 1
Late RT Toxicity: Skin: NOS (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension NOS (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAS x 8 Weeks (N=747) | TAS x 28 Weeks (N=735)
Constipation (Gastrointestinal disorders) | 25 | 42
Diarrhea NOS (Gastrointestinal disorders) | 238 | 245
Late RT Toxicity: Other GI: NOS (Gastrointestinal disorders) | 135 | 159
Late RT Toxicity: Small/Large Intestine: NOS (Gastrointestinal disorders) | 194 | 196
Proctitis NOS (Gastrointestinal disorders) | 173 | 164
Late RT Toxicity: Other: NOS (General disorders) | 113 | 124
Fatigue (General disorders) | 159 | 224
Dermatitis radiation NOS (Injury, poisoning and procedural complications) | 103 | 89
Alanine aminotransferase increased (Investigations) | 92 | 104
Blood bilirubin increased (Investigations) | 30 | 41
Libido decreased (Psychiatric disorders) | 17 | 51
Dysuria (Renal and urinary disorders) | 82 | 85
Late RT Toxicity: Bladder: NOS (Renal and urinary disorders) | 260 | 270
Urinary frequency (Renal and urinary disorders) | 444 | 456
Gynaecomastia (Reproductive system and breast disorders) | 34 | 107
Impotence (Reproductive system and breast disorders) | 64 | 132
Late RT Toxicity: Other GU: NOS (Reproductive system and breast disorders) | 191 | 194
Menopausal symptoms (Vascular disorders) | 458 | 596

LIMITATIONS AND CAVEATS:
The data monitoring committee decided in June 2012 after the first interim analysis that the trial should be reported early due to the low number of events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.